CLINICAL TRIAL: NCT05042674
Title: Clinical Study on Rapid Antioxidant Protection and Immune Modulating Effects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Principal Investigator, Gitte Jensen, Ph.D., Research Director, Natural Immune Systems Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NIS174-003
Record Dates: First submitted 2021-09-04; First posted 2021-09-13 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Ergothioneine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Placebo, Ergothioneine 25mg, Ergothioneine 25mg for 1 week daily (Other): Participants will consume placebo on first study day, consume 25mg of ergothioneine on second study day, then consume 25mg of ergothioneine daily for 1 week
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Ergothioneine, 25 miligrams; Dietary Supplement: Ergothioneine, 25 miligrams, daily for 1 week

INTERVENTIONS:
Dietary Supplement: Placebo — after a blood draw placebo will be consumed followed by 2 additional blood draws
Dietary Supplement: Ergothioneine, 25 miligrams — after a blood draw 25 miligrams of ergothioneine will be consumed followed be 2 additional blood draws
Dietary Supplement: Ergothioneine, 25 miligrams, daily for 1 week — a blood draw will be administered after a week of consuming 25mg ergothioneine daily

SUMMARY:
A trial on acute antioxidant protection and immune effects when 24 people consume a novel nutraceutical blend compared to a placebo on different test days.

DETAILED DESCRIPTION:
A randomized, cross-over study design will be used to evaluate immune effects of consumption of 25 mg ergothioneine. On the first clinic day, participants will take a placebo with a one week wash out. Following the wash out week, participants will take 25 mg ergothioneine for 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Willing to comply with a 24-hour wash-out period for vitamins and nutritional supplements
* Willing to maintain a consistent diet and lifestyle routine throughout the study
* Willing to avoid consumption of meals where the predominant ingredients include mushrooms, seafood, and organ meat (liver, heart).*
* Willing to abstaining from exercising on the morning of a study visit
* Willing to abstain from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit
* Willing to abstain from music, candy, gum, computer/cell phone use, during clinic visits.

Exclusion Criteria:

* Previous major gastrointestinal surgery
* Active chronic immunological disease
* Currently taking daily OTC medications, prescription pain medications, antipsychotic medications, anti-inflammatory nutritional supplements judged by the study coordinator to negate or camouflage the effects if the test product, nutritional supplements containing medicinal mushroom extracts
* Diagnose with Type I diabetes, autoimmune disorders
* Getting regular joint injections
* Active severe chronic disease (such as HIV, chronic hepatitis)
* Currently experiencing intense stressful events/ life changes
* Currently in intensive athletic training
* Experiencing an unusual sleep routine
* Unwilling to maintain a constant intake of supplements over the duration of the study
* Anxiety about having blood drawn
* Women who are pregnant, nursing, or trying to become pregnant
* Known food allergies to ingredients in test product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-03-25 (Estimated); Study Completion 2023-05-05 (Estimated)

PRIMARY OUTCOMES:
Change in level of reduced glutathione | 2 hours
  Mean fluorescence

SECONDARY OUTCOMES:
Change in mitochondrial mass and mitochondrial potential from baseline | 2 hours
  Mean fluorescence

OTHER OUTCOMES:
Change in level of reduced glutathione | 1 week
  Mean fluorescence
Change in mitochondrial mass and mitochondrial potential from baseline | 1 week
  Mean fluorescence

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Jensen, PhD, Principal Investigator — NIS Labs
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No